CLINICAL TRIAL: NCT02372942
Title: Lactoferrin or Progesterone for Prevention of Preterm Delivery
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Padova (Other)
Responsible Party: Principal Investigator, Erich Cosmi MD, PhD, Associate Professor in Obstetrica and Gynecolgy, University of Padova
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: University of Padua
Record Dates: First submitted 2015-02-07; First posted 2015-02-26 (Estimated); Last update posted 2018-05-08 (Actual); Status verified 2018-05

CONDITIONS: Preterm Delivery
Keywords: efficacy; prevention
MeSH Terms: conditions — Premature Birth | interventions — Progesterone

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Lattoferrin (Experimental): Use of Lattoferin for prevention of preterm delivery
  Interventions: Drug: Lattoferrin
- Progesterone (Experimental): Use of Progesterone for prevention of preterm delivery
  Interventions: Drug: Progesterone

INTERVENTIONS:
Drug: Lattoferrin — 515 pregnant women using lattoferrin to prevent preterm delivery
  Other Names: Difesan
  Arms: Lattoferrin
Drug: Progesterone — 515 pregnant women using lattofferrin to preventf preterm delivery lattoferrin or progesterone
  Other Names: Progeffik
  Arms: Progesterone

SUMMARY:
Primary endpoint will be evaluate the effectiveness of vaginal lactoferrin in the reduction of the 30% of preterm deliveries versus the use of progesterone, in specific selected patients, with consequent improvement in neonatal outcome.

Secondary endpoint will be compare antibacterial and anti-inflammatory activity of lactoferrin by evaluation of systemic biochemical and urinary markers.

DETAILED DESCRIPTION:
AIM OF THE STUDY Primary endpoint will be evaluate the effectiveness of vaginal lactoferrin in the reduction of the 30% of preterm deliveries versus the use of progesterone, in specific selected patients, with consequent improvement in neonatal outcome.

Secondary endpoint will be compare antibacterial and anti-inflammatory activity of lactoferrin by evaluation of systemic biochemical and urinary markers.

MATHERIAL AND METHODS Type of study: This is a randomized and open-label study (lactoferrin vs progesterone), multicenter.

Population of study: pregnant women 18-43 years aged with singleton pregnancy, between 24 and 34 weeks' gestation, who were at risk of preterm delivery.

Investigational products:

* Lactoferrin (Difesan, vaginal tablets 300 mg); it is used in acute vaginosis (300 mg intravaginally once a day for seven consecutives days). Since there are no side effects, for experimental purpose it will be used until 34 weeks of gestation.
* Progesterone (Progeffik, vaginal suppositories 200 mg); in case of risk of premature delivery the treatment consist in 200 mg intravaginally once a day, for a maximum of 10 weeks. In this protocol it will be used until 34 weeks of gestation.

Duration of study: considering the prevalence of the disease and the number of deliveries for years, it will be concluded in 2015.

Centers: Department of Women's and Child's Health, Obstetrics and Gynecology Clinic, University of Padua, Italy.

Others: Udine, Italy "S. Maria della Misericordia Hospital" Vicenza, Italy "S. Bortolo Hospital" Ferrara, Italy Bologna, Italy Treviso, Italy

Inclusion criteria:

* cervical length less than 25 mm between 24 and 34 weeks' gestation (with or without funnelling)
* cervical effacement less than 50 percent and cervical dilatation less than 3 cm
* uterine contractions less than 4 in 30 minutes
* singleton pregnancy
* absence of chorioamnionitis signs (white cells count< 15.000, Reactive Protein C< 10 mg/l, Procalcitonin levels < 0,05 ng/ml),
* absence of premature membrane rupture (pPROM).

Exclusion criteria:

1. Fetal abnormalities such as severe intrauterine growth restriction and fetal malformations with progressive deterioration
2. Maternal diseases such as gestation diabetes insulin-treated, severe nephropaties, severe cardiopathies, autoimmune diseases
3. Twin pregnancy
4. Signs of maternal infections (chorioamnionitis)
5. Premature rupture of membrane

Previous progesterone therapy during first trimester is not a contraindication for the inclusion of the patients (interval at least 8-10 weeks of gestation).

Previous preterm birth is not a exclusion criteria for the randomization.

Evaluation scheme:

1. Verification of maternal compatibility with study criteria.
2. Accurate personal, familiar and obstetrical anamnesis.
3. Management of the patient according to the clinical protocol in case of risk of premature delivery (induction of fetal lung maturity and tocolitic therapy)
4. Informed consent.
5. Patient randomization.
6. Obstetrical and ultrasound evaluation of pregnancy (cervical length, fetal growth and fetal well-being at 7, 15 and 30 days from the randomized).
7. Monitoring of inflammatory markers (white blood cells, reactive protein C and procalcitonin) at diagnosis, at 7 and 15 days from the recovery.
8. Execution of vaginal swab and urine culture at diagnosis and at 30 days from the recovery.
9. Registration of pregnancy data, delivery and neonatal out come.

EXCLUSION CRITERIA

The patient will be excluded from the study if they do occur the following conditions during administration of lactoferrin or progesterone:

1. Presence of regular, painful and frequent uterine contractions and progressive change in the cervix (cervical effacement of 80 percent or greater and cervical dilatation greater than 3 cm)
2. Modification of the inflammatory markers that are associated to changes to the obstetrical visit or cervical length.

There are no costs because the check-up expected for the patient belong to clinic routine.

The patients will not pay the treatment because it will be provided by the Principal Investigator.

MEASUREMENT

1. Obstetrical data: during recovery and till delivery (course of pregnancy, sonography examination, biochemical tests, complications.
2. Perinatal data: gestational age at the time of delivery, way of delivery, sex, weight, Apgar score, arterial and venous ph, base excess, p02, days of recovery in neonatal intensive care unit, mechanical ventilation, neonatal morbidity, breastfeeding.
3. Epidemiological data: maternal and paternal data (age, BMI, smoke and socio-economical status, parity, ethnic group, personal history). Familiar history.

SAMPLE SIZE The patients enrolled in the study are those treated for high risk of preterm delivery that respected inclusion criteria. They are randomized in two groups, one group is submitted to lactofferin, the other group receives progesterone. For the calculation of sample size we considered a recent review that concluded that progesterone treatment decreased the median risk of preterm birth by 22% (Likis F et al. Progestogens for preterm birth prevention. Obstet Gynecol October 2012).

The primary outcome is to show that lactoferrin decreases the median risk of preterm birth by 30% ; We considered alfa 5% and predictive value of 80%; considering 10% of drop out we will randomize 1030 women.

[n=p1(p1-100)+p2(p2-100)/(p1-p2)2 x 7.9]

ELIGIBILITY:
Inclusion Criteria:

* Cervical length less than 25 mm between 24 and 34 weeks' gestation (with or without funnelling)

  * cervical effacement less than 50 percent and cervical dilatation less than 3 cm
  * uterine contractions less than 4 in 30 minutes
  * singleton pregnancy
  * absence of chorioamnionitis signs (white cells count< 15.000, Reactive Protein C< 10 mg/l, Procalcitonin levels < 0,05 ng/ml),
  * absence of premature membrane rupture (pPROM).

Exclusion Criteria:

* Fetal abnormalities such as severe intrauterine growth restriction and fetal malformations with progressive deterioration
* Maternal diseases such as gestation diabetes insulin-treated, severe nephropaties, severe cardiopathies, autoimmune diseases
* Twin pregnancy
* Signs of maternal infections (chorioamnionitis)
* Premature rupture of membrane

Ages: 18 Years to 43 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 1030 (Estimated)
Dates: Start 2014-02 (Actual); Primary Completion 2019-11 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
delayed days of birth using lattoferrin or progesterone | days or weeks

SECONDARY OUTCOMES:
neonatal outcome | 28 days and 2 years follou-up

CONTACTS AND LOCATIONS:
Overall Officials: Erich Cosmi, MD, PhD, Principal Investigator — University of Padova
Locations (1):
- University of Padua, Padua, Italy

IPD SHARING:
Plan to Share IPD: Yes